CLINICAL TRIAL: NCT01294124
Title: Investigating The Neurobiology of Tinnitus
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: NMCSD.2013.0021; CDMRP (Other Grant/Funding Number: DM102565)
Record Dates: First submitted 2011-02-09; First posted 2011-02-11 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Tinnitus; Traumatic Brain Injury; Post Traumatic Stress Disorder
MeSH Terms: conditions — Tinnitus; Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- No Tinnitus: The absence of tinnitus will be based on the participants' responses to questions 8a, 9c, and 9d of the Post-Deployment Health Assessment (PDHA).
- Tinnitus: The presence of tinnitus will be based on the participants' responses to questions 8a, 9c, and 9d of the Post-Deployment Health Assessment (PDHA).

SUMMARY:
The investigators hypothesize that individual differences exist in resting-state cortical attention, control, sensory, and emotion networks prior to noise exposure and these differences predispose some to the development of bothersome tinnitus. Furthermore, the investigators hypothesize that these changes in functional connectivity of these vulnerable systems after noise exposure are responsible for tinnitus. The proposed study will use a case-control cohort study design. Cases will be those soldiers who develop tinnitus and controls will be those who do not. This will be the first prospective study of tinnitus and will provide important information about the neurobiology of tinnitus.

If a cortical neural network etiology for bothersome tinnitus is confirmed, it will be an astounding, powerful, paradigm shifting model for the diagnosis, prevention and, most importantly, treatment of tinnitus. Furthermore, if a battery of neurocognitive tests can identify soldiers at risk for the development of tinnitus then appropriate primary prevention strategies can be introduced.

There are three Specific Aims to this project.

Specific Aim 1. To determine if soldiers who develop tinnitus display pre-deployment differences in a set of physical, functional, cognitive, vulnerability, perpetuating factors, pre-deployment neurocognitive scores, or neuroimaging features compared to soldiers who do not develop tinnitus ("control group").

Specific Aim 2. To determine if particular scores on neurocognitive tests or neuroimaging features of functional/structural connectivity networks are associated with the development of tinnitus.

Specific Aim 3. To identify a set of pre-deployment physical, functional, cognitive, vulnerability, and perpetuating factors, neurocognitive responses, and neuroimaging features that are associated with the development of tinnitus.

The investigators plan to recruit 200 soldiers, between the ages of 18 and 30 years who do not have hearing loss or tinnitus and have never been deployed to military theater. The soldier participants will undergo a variety of tests before and after deployment, which will include a hearing test, neurocognitive tests (i.e., brain function tests), and a variety of novel radiologic imaging studies of the brain. One of these novel radiologic imaging studies is functional connectivity Magnetic Resonance Imaging, a proven methodology that monitors changes in brain activity and connections based on blood flow between different brain areas and levels of consumption of oxygen. This information is used to describe the condition of important neural networks responsible for such things as attention, mood, sensation, vision, hearing, and introspection or self-contemplation.

ELIGIBILITY:
Inclusion Criteria:

* Active duty or reserve military personnel with MOS job code 11B, 11C, 19D, or 19K
* Men and women between the ages of 18 and 30 years
* Scheduled for first deployment to military theater
* Must be able to read, write, and understand English
* Willing to sign Request Pertaining to Military Records (Form 180) to allow study personnel to access medical records for the purposes of this study.

Exclusion Criteria:

* History of hearing loss or tinnitus
* Currently taking medication for depression, anxiety, or other DSM IV Axis 1 disorder
* History of head trauma sufficient to cause loss of consciousness for 30 minutes or greater
* History of surgery to the brain
* History of claustrophobia
* Presence of metallic implants in the head and upper cervical region that are non-MRI compatible and would prohibit use of MRI.
* At any time in the past, prior deployment or employment in military theater
* Currently pregnant

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Active-duty or reserve United States military personnel between the ages of 18 and 30 of either sex, all races and ethnicity, who are scheduled for initial deployment to theater with a Military Occupational Specialty code (MOS) of 11B Infantryman, 11C Indirect Fire Infantryman, 19D Calvary Scout, or 19K Armor Crewman.
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Development of Tinnitus | Post-deployment assessment will occur no sooner than 90 days from return from active military theater.
  The presence of tinnitus will be based on the participants' responses to questions 8a, 9c, and 9d of the Post-Deployment Health Assessment (PDHA).

SECONDARY OUTCOMES:
Mild Traumatic Brain Injury | Post-deployment assessment will occur no sooner than 90 days from return from active military theater.
  Mild Traumatic Brain Injury - Ohio State University TBI Identification Method (OSU TBI-ID version 12-10-08)(Corrigan and Bogner 2007)
Post Traumatic Stress Disorder | Post-deployment assessment will occur no sooner than 90 days from return from active military theater.
  Subjects whose military medical record or PDHA suggests PTSD will be asked to complete the Clinician Administered PTSD Scale (CAPS).(Blake et al. 1995; Weathers and Litz 1994)

CONTACTS AND LOCATIONS:
Overall Officials: Jay F. Piccirillo, MD, Principal Investigator — Washington University School of Medicine; Sean Wise, CAPT., M.D., Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center, San Diego, California, United States